CLINICAL TRIAL: NCT05634343
Title: Laughter Therapy and Mindfulness Practices in Nurses
Brief Title: Laughter Therapy and Mindfulness Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagihan Koroglu Kaba (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Nagihan Koroglu Kaba, Lecturer, Bayburt University
Organization: Bayburt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NKOROGLUKABA-TEZ-KTÜ
Record Dates: First submitted 2022-11-18; First posted 2022-12-02 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Nurse's Role
Keywords: Mindfulness, Attention, Laughter therapy, Job performance, Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: The research examines the effects of laughter and mindfulness on some parameters (fatigue, performance and attention) in nurses.
Who Masked: Participant, Investigator
Masking Description: Simple random numbers table was used to determine the nurses to be sampled. 673 nurses working in KTU Farabi Hospital were listed and numbered, and the starting point was chosen from the random numbers table, followed by the columns downwards, and the sample number was reached. If the sample could not be reached due to reasons such as the criteria were not met or the research invitation was not accepted, the sample selection was continued from the random numbers table until the sample number was reached. Then, in order to create homogeneous groups in the assignment of nurses to the experimental and control groups, equal numbers of triple groups were formed by matching according to the unit/service (internal, surgical, specialized unit) and professional experience (10 years and below, 11 years and above).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group 1 (Experimental): The laughter therapy program consists of 16 sessions, twice a week for eight weeks. Each session; It is planned to last 30-45 minutes with a maximum of 25 nurses.
  Interventions: Other: experimental group 1
- experimental group 2 (Experimental): The mindfulness practice program consists of 16 sessions, twice a week for eight weeks. Each session is planned to last 45-60 minutes with a maximum of 25 nurses.
  Interventions: Other: experimantal group 2
- Control Group (No Intervention): No intervention was made in the control group.

INTERVENTIONS:
Other: experimental group 1 — Laughter therapy, also called therapeutic laughter, is used to relieve pain and stress and to promote a general sense of well-being. Laughter therapy is simply a method of 'laughing for no reason' in which the person interacts in a group setting with improvisation or pantomime-like exercises and childish games without humour, jokes or funny events. The aim is thus to benefit from laughter.
  Arms: experimental group 1
Other: experimantal group 2 — Mindfulness is purposefully drawing attention in the desired direction so that we can stay in the present moment without judgment. It is also defined as a conscious understanding of what is happening in the moment we live in with an open and loving attitude. According to another definition, mindfulness includes paying attention to what is happening in the present moment, noticing the quality of this attention, and accepting what is noticed without judgment. With conscious awareness, the individual discovers how to live in harmony with all the events that take place in the present moment, place and time, without any evaluation, rather than the sorrows and regrets of the past, the anxieties and worries of the future. Mindfulness helps us to relate to our experiences by enabling us to see the positive-negative, good-bad experiences we have had objectively.
  Arms: experimental group 2

SUMMARY:
Nurses working by shifts under intense stress and pressure and using complicated technological products- undergo fatigue and attention deficit with the effect of the many negative factors caused by work setting. This threatens patient and staff safety as well as leads to communicational problems, work absenteeism, lowered motivation, inability to control stress and poor work performance and productivity among nurses as well. In this sense; laughter therapy and mindfulness practices may help nurses cope with these problems because some experimental studies proved that both methods showed many benefits in different samples. However; no studies in which these two methods were compared among nurses were encountered. Therefore; the study -being in experimental design and randomized controlled trial- will be undertaken with a total of 111 nurses employed at a university hospital -37 nurses allocated to the experimental 1 group, 37 nurses to the experimental 2 group and 37 nurses to the control group-. First; Computer-Based Sustained Attention Test, the Stroop Test Çapa Version, The Chalder Fatigue Scale (CFQ) and Individual Work Performance Questionnaire will be administered to the nurses of the experimental and control groups as a pre-test. Then; nurses of the experimental 1 group will join sessions of laughter therapy (30-45 minutes twice a week for 8 weeks) and nurses of the experimental 2 group will join sessions of mindfulness practices (45-60 minutes twice a week for 8 weeks) for two months. One month later when the sessions are started, a mid test will be administered and soon after the sessions are completed a post test will be administered to the nurses via Computer-Based Sustained Attention Test, the Stroop Test Çapa Version, The Chalder Fatigue Scale (CFQ) and Individual Work Performance Questionnaire. One month later after the post test; a follow-up will be performed using the same tools. As a result; the effects of both applications on fatigue, attention and performance will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* at least 6 months experience
* volunteering
* alternative work schedule

Exclusion Criteria:

* Not being a nurse,
* Pregnancy
* Diagnosis of colour blindness, cardiovascular, psychological diseases
* Meditating before

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | First day
  This form developed by the researcher consists of six questions about the characteristics of nurses.
Chalder Fatigue Scale | First day
  The scale was developed in 1993 to measure the severity of fatigue. The scale has two sub-dimensions (physical and mental) and consists of 11 items. The total fatigue score is obtained by summing the scores of all items. Higher scores indicate greater severity of fatigue.
Computer-Based Sustainable Attention Test | First day
  Developed in 2006, the test measures sustained attention at three levels: easy, medium and difficult. A minimum of 0 and a maximum of 10 are taken from each level. An increase in the test score indicates an increase in the level of sustained attention.
Stroop Test Çapa Form | First day
  The Stroop form developed by Weintraub in 2000 was adapted to Turkish by Emek Savaş et al. The test is used to determine the selective attention and reaction time of individuals. In the test, there are two stimulus cards and a total of 60 items placed on each card in the order of 6 x 10. The first card contains small rectangles of red, green and blue, while the second card has color names written in mismatched ink colors. The Stroop test is one of the most frequently used tests in neuropsychological evaluation. The fact that it can be applied to people of all age groups in a short time increases the preferability of the test.
Individual Job Performance Scale | First day
  The scale developed by Koopmans et al. in 2013 measures employee performance in three dimensions (task, contextual, counterproductive behaviour). The scale has 14 items and is a five-point Likert scale.

SECONDARY OUTCOMES:
Chalder Fatigue Scale | At the end of the 1st month
  The scale was developed in 1993 to measure the severity of fatigue. The scale has two sub-dimensions (physical and mental) and consists of 11 items. The total fatigue score is obtained by summing the scores of all items. Higher scores indicate greater severity of fatigue.
Computer-Based Sustainable Attention Test | At the end of the 1st month
  Developed in 2006, the test measures sustained attention at three levels: easy, medium and difficult. A minimum of 0 and a maximum of 10 are taken from each level. An increase in the test score indicates an increase in the level of sustained attention.
Stroop Test Çapa Form | At the end of the 1st month
  The Stroop form developed by Weintraub in 2000 was adapted to Turkish by Emek Savaş et al. The test is used to determine the selective attention and reaction time of individuals. In the test, there are two stimulus cards and a total of 60 items placed on each card in the order of 6 x 10. The first card contains small rectangles of red, green and blue, while the second card has color names written in mismatched ink colors. The Stroop test is one of the most frequently used tests in neuropsychological evaluation. The fact that it can be applied to people of all age groups in a short time increases the preferability of the test.
Individual Job Performance Scale | At the end of the 1st month
  The scale developed by Koopmans et al. in 2013 measures employee performance in three dimensions (task, contextual, counterproductive behaviour). The scale has 14 items and is a five-point Likert scale.
Chalder Fatigue Scale | At the end of the 2st month
  The scale was developed in 1993 to measure the severity of fatigue. The scale has two sub-dimensions (physical and mental) and consists of 11 items. The total fatigue score is obtained by summing the scores of all items. Higher scores indicate greater severity of fatigue.
Computer-Based Sustainable Attention Test | At the end of the 2st month
  Developed in 2006, the test measures sustained attention at three levels: easy, medium and difficult. A minimum of 0 and a maximum of 10 are taken from each level. An increase in the test score indicates an increase in the level of sustained attention.
Stroop Test Çapa Form | At the end of the 2st month
  The Stroop form developed by Weintraub in 2000 was adapted to Turkish by Emek Savaş et al. The test is used to determine the selective attention and reaction time of individuals. In the test, there are two stimulus cards and a total of 60 items placed on each card in the order of 6 x 10. The first card contains small rectangles of red, green and blue, while the second card has color names written in mismatched ink colors. The Stroop test is one of the most frequently used tests in neuropsychological evaluation. The fact that it can be applied to people of all age groups in a short time increases the preferability of the test.
Individual Job Performance Scale | At the end of the 2st month
  The scale developed by Koopmans et al. in 2013 measures employee performance in three dimensions (task, contextual, counterproductive behaviour). The scale has 14 items and is a five-point Likert scale.
Chalder Fatigue Scale | At the end of the 3st month
  The scale was developed in 1993 to measure the severity of fatigue. The scale has two sub-dimensions (physical and mental) and consists of 11 items. The total fatigue score is obtained by summing the scores of all items. Higher scores indicate greater severity of fatigue.
Computer-Based Sustainable Attention Test | At the end of the 3st month
  Developed in 2006, the test measures sustained attention at three levels: easy, medium and difficult. A minimum of 0 and a maximum of 10 are taken from each level. An increase in the test score indicates an increase in the level of sustained attention.
Stroop Test Çapa Form | At the end of the 3st month
  The Stroop form developed by Weintraub in 2000 was adapted to Turkish by Emek Savaş et al. The test is used to determine the selective attention and reaction time of individuals. In the test, there are two stimulus cards and a total of 60 items placed on each card in the order of 6 x 10. The first card contains small rectangles of red, green and blue, while the second card has color names written in mismatched ink colors. The Stroop test is one of the most frequently used tests in neuropsychological evaluation. The fact that it can be applied to people of all age groups in a short time increases the preferability of the test.
Individual Job Performance Scale | At the end of the 3st month
  The scale developed by Koopmans et al. in 2013 measures employee performance in three dimensions (task, contextual, counterproductive behaviour). The scale has 14 items and is a five-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayburt University, Bayburt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koroglu Kaba N, Ozturk H. The Effects of Laughter Yoga and Mindfulness on Nurses' Fatigue, Work Performance and Attention Levels: A Randomized Controlled Study. Clin Nurse Spec. 2025 Nov-Dec 01;39(6):260-268. doi: 10.1097/NUR.0000000000000927. PMID 41118502